CLINICAL TRIAL: NCT00065429
Title: A Phase I, Open-Label, Dose Escalation Study of Weekly Dosing With BB-10901, Followed by a Phase II Efficacy Expansion
Brief Title: Safety Study Using Weekly Infusions of BB-10901 in Patients With Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ImmunoGen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C10/IVB/001; NCT00074256 (obsolete NCT alias)
Record Dates: First submitted 2003-07-23; First posted 2003-07-24 (Estimated); Results first posted 2012-06-20 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — lorvotuzumab mertansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- BB-10901, 5mg/m2 - Phase I (Experimental)
  Interventions: Drug: BB-10901
- BB-10901, 10 mg/m2 - Phase I (Experimental)
  Interventions: Drug: BB-10901
- BB-10901, 20 mg/m2 - Phase I (Experimental)
  Interventions: Drug: BB-10901
- BB-10901, 40 mg/m2 - Phase I (Experimental)
  Interventions: Drug: BB-10901
- BB-10901, 60 mg/m2 - Phase I & Phase II (Experimental): Phase I and Phase II were consecutive and sequential. Different patients received the 60mg/m2 dose in Phase I and in Phase II.
  Interventions: Drug: BB-10901
- BB-10901, 67.5 mg/m2 - Phase I (Experimental)
  Interventions: Drug: BB-10901
- BB-10901, 75 mg/m2 - Phase I (Experimental)
  Interventions: Drug: BB-10901

INTERVENTIONS:
Drug: BB-10901 — I.V. Infusion - See "Arms" for dosage - Once/Week for three weeks - Until Progression of disease.

SUMMARY:
This study was a Phase I/II trial primarily focused on efficacy of BB-10901 in relapsed small cell lung cancer and other solid tumors.

DETAILED DESCRIPTION:
The Phase II efficacy expansion was restricted to SCLC patients with relapsed disease and the MTD was determined by the Phase I portion of the trial (60mg/m2).

ELIGIBILITY:
Inclusion:

* Histologically or Cytologically proven SCLC, CD 56+ small cell carcinoma of unknown origin, or CD56+ non-pulmonary small cell carcinoma
* Relapsed disease; defined as patients with an initial response (partial or complete) to first-line therapy, then relapse more than 3 months after completion of last chemotherapy.
* Patients must have received no more than 3 prior chemotherapy regimen.
* Patients must have measurable disease defined as: Lesions that can be measured in at least one dimension according to RECIST
* Predicted survival of 3 months or more
* Zubrod performance status 0-2
* Patients must not have received chemotherapy or radiation therapy within 4 weeks of study entry, nor have planned surgery.
* Absolute neutrophils greater than or equal to 1.5 x 10^9/l, hemoglobin greater than or equal to 9g/dl and platelets greater than or equal to 100 x 10^9/l.
* Creatinine less than or equal to 1.5 times the upper limit of normal
* AST/ALT less than or equal to 3 times the upper limit of normal without liver metastases; less than or equal to 5 times the upper limit of normal with liver metastases and bilirubin less than or equal to 1.5 times the upper limit of normal.
* Patients must have normal thyroid function (patients receiving thyroxin replacement therapy who are biochemically euthyroid may be enrolled).
* Women of childbearing potential must provide a negative pregnancy test at screening and use adequate contraception in the opinion of the investigator, for the duration of study.
* Patients must be capable of understanding the nature of the trial and must give written witnessed informed consent prior to any screening procedure.

Exclusion:

* Significant residual neurological or cardiac toxicity (grade 3 or 4) following previous chemotherapy
* Patients who are concurrently receiving other anti-neoplastic treatment (chemotherapy, radiotherapy, or immunotherapy including steroid therapy).
* Myocardial infarction within 6 months of study entry, unstable angina pectoris, uncontrolled congestive heart failure, uncontrolled arrythmia, severe aortic stenosis, a history of multiple sclerosis, or other demyelinating disease, Eaton-Lambert Syndrome, history of hemorrhagic stroke, any CNS injury with residual neurologic deficit, ischaemic stroke within the last 6 months, current known herpes zoster (shingles), or cytomegalovirus infection, or a history of recurrent infections with these viruses, chronic alcoholism, serious concomitant infection, or any other concomitant illness considered significant enough to interfere with the study outcome.
* Other investigational agents must not be taken during the study or within 4 weeks of study entry.
* Previous monoclonal antibody therapy
* Patients must not have known central nervous system metastases
* Previous malignancy with < 5 year disease free interval from the last therapeutic intervention, except for adequately treated basal cell carcinoma of the skin or carcinoma in situ of the cervix.
* Patient unwilling or unable to tolerate and comply with the requirements of the study.
* Pregnant or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2003-04; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Cancer Center of Florida, Ocoee, Florida
  - Baystate Medical Center, Springfield, Massachusetts
  - New York Oncology Hematology, Albany, New York
  - The Ohio State University, Colombus, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Northwest Cancer Specialists, Vancouver, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In Phase I, 32 patients were treated with doses ranging from 5 mg/m2/week to 75 mg/m2/week, with 9 patients treated at the MTD dose of 60 mg/m2/week. In Phase II, 32 advanced cancer patients were treated with BB-10901 at a dose of 60 mg/m2/week. (Total N=64)
Pre-assignment Details: This study was an open-label study. All patients that consented to the trial and met inclusion/exclusion criteria were enrolled.
Groups:
- IMGN 5 mg/m2: Arm 1, Phase 1
- IMGN 10 mg/m2: Arm 2, Phase 1
- IMGN 20 mg/m2: Arm 3, Phase 1
- IMGN 40 mg/m2: Arm 4, Phase 1
- IMGN 60 mg/m2: Arm 5, Phase 1 and 2
- IMGN 67.5 mg/m2: Arm 6, Phase 1
- IMGN 75 mg/m2: Arm 7, Phase 1
Period: Phase I - May 2001 - Oct 2002
Arm/Group | IMGN 5 mg/m2 | IMGN 10 mg/m2 | IMGN 20 mg/m2 | IMGN 40 mg/m2 | IMGN 60 mg/m2 | IMGN 67.5 mg/m2 | IMGN 75 mg/m2
Started | 4 | 3 | 4 | 4 | 9 | 4 | 4
Completed | 3 | 3 | 3 | 3 | 8 | 2 | 2
Not Completed | 1 | 0 | 1 | 1 | 1 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 1 | 2
Period: Phase II - Apr 2003 - Aug 2008
Arm/Group | IMGN 5 mg/m2 | IMGN 10 mg/m2 | IMGN 20 mg/m2 | IMGN 40 mg/m2 | IMGN 60 mg/m2 | IMGN 67.5 mg/m2 | IMGN 75 mg/m2
Started | 0 (Patients participated at this dose level only in Phase 1.) | 0 (Patients participated at this dose level only in Phase 1.) | 0 (Patients participated at this dose level only in Phase 1.) | 0 (Patients participated at this dose level only in Phase 1.) | 32 (All 32 patients enrolled in Phase 2 were at 60 mg/m2.) | 0 (Patients participated at this dose level only in Phase 1.) | 0 (Patients participated at this dose level only in Phase 1.)
Completed | 0 | 0 | 0 | 0 | 26 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 6 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 4 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IMGN 5 mg/m2 | IMGN 10 mg/m2 | IMGN 20 mg/m2 | IMGN 40 mg/m2 | IMGN 60 mg/m2 | IMGN 67.5 mg/m2 | IMGN 75 mg/m2 | Total
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 41 | 4 | 4 | 64
Age Continuous [Mean (Standard Deviation); unit: years] | 64.0 (10.86) | 59.0 (13.08) | 60.0 (12.65) | 59.8 (9.07) | 61.2 (10.1) | 59.5 (4.8) | 54.5 (9.5) | 62.67 (10.01)
Age, Customized [Number; unit: participants]
  >=18 years | 4 | 3 | 4 | 4 | 41 | 4 | 4 | 64
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 1 | 14 | 1 | 4 | 23
  Male | 4 | 2 | 2 | 3 | 27 | 3 | 0 | 41
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 4 | 4 | 41 | 4 | 4 | 64

OUTCOME MEASURES:

1. Primary Outcome: Phase I Toxicity Based Upon Adverse Events Clasified by the NCI Common Terminology Ctireria Version 2.0 (Phase I)
Description: Dose limiting toxicities graded according to common terminology criteria for advers events, version 2.0 and defined as AEs (probably/definitely related to study drug) meeting the NCI CTC criteria, assessed on the basis of the first cycle of therapy (4 weeks of weekly dosing/2 week fu): Hematologic Tox (Grade 4 neutropenia ≥ 5 days, Grade 4 thrombocytopenia, neutropenic infection); Non-Hem Toxicity: (Any grade 3 or 4 non-hematologic toxicity, excluding nausea, vomiting, diarrhea and alopecia); Toxicity present at Screening (concurrent conditions), an increase in severity of 2 or more grades.
Time Frame: every 6 weeks
Population: All Phase I enrolled patients who received study drug were analyzed for DLTs.
Measure: Number; unit: participants
Groups:
- Phase I: The study had a conventional open-label cytotoxic study design to determine the safety, tolerability and MTD, preliminary efficacy signal and PK. Once the MTD was found in Phase I, the study would continue to a Phase II expansion at the MTD and the MTD-1 dose levels determined in Phase I. Infusions given at 1-week intervals were expected to provide intermittent exposure with no accumulation of BB-10901. The maximum duration of treatment at each dose level was 4 cycles of treatment; patients with evidence of response were eligible to continue for up to 6 cycles of treatment. Dose levels planned were 5, 10, 20, 40, 60 and 90 mg/m2/week. Three patients were to be enrolled per dose level with dose escalation when 1 of 3 patients completed 1 cycle and 2 patients had received at least 2 weekly infusions and were eligible for their third infusion, all without DLT. Once the MTD had been defined, 3 more patients were planned for enrollment at the MTD and 3 patients at the MTD-1 level.
Arm/Group | Phase I
Number analyzed (Participants) | 32
participants
  Non-infective meningitis | 3 (0) [0 to 5]
  Hyperesthesia Grade 4 | 1
  Peripheral sensory neuropathy Grade 3 | 1
  Fatigue Grade 3 | 1
  Headache Grade 3 | 1

2. Primary Outcome: Response Evaluation Criteria in Solid Tumors (RESIST) [Phase I and II]
Description: Response was evaluated by RESIST and Investigator assessment at baseline and every 6 weeks. CR: all target lesions disappear with no clinical or radiographic evidence of disease progression in 2 observations. PR: At least 30% decrease in sum of the longest diameters of target lesions shown in 2 observations. SD: does not qalify for PR or PD based on 2 observations. PD: Either a) the appearance of one or more new lesions, or b) at least a 20% increase in the sum of longest diameters of target lesions
Time Frame: 6 weeks
Population: All patients with a baseline and follow up imaging scan were evaluated. Data represents information following the first cycle of treatment.
Measure: Number; unit: participants
Groups:
- Phase II: For Phase II, the planned design was to use a Gehan's two-stage design [4], with a total of 14 patients assigned to each of 2 dose levels. The dose levels to be tested were to be selected after review of the Phase I data and, assuming evidence of efficacy was seen in that phase, were likely to be the MTD and MTD-1.
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 29 | 29
participants
  Complete Response (CR) or Partial Response (PR) | 0 | 2
  Stable Disease | 10 | 10
  Progressive Disease (PD) | 16 | 17
  Unknown | 3 | 0

ADVERSE EVENTS:
Time Frame: From 29 May, 2001 to 16 Oct, 2008
Arm/Group | IMGN 5 mg/m2 | IMGN 10 mg/m2 | IMGN 20 mg/m2 | IMGN 40 mg/m2 | IMGN 60 mg/m2 | IMGN 67.5 mg/m2 | IMGN 75 mg/m2
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/3 | 0/4 | 1/4 | 5/41 | 1/4 | 0/4
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 3/4 | 4/4 | 41/41 | 4/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMGN 5 mg/m2 (N=4) | IMGN 10 mg/m2 (N=3) | IMGN 20 mg/m2 (N=4) | IMGN 40 mg/m2 (N=4) | IMGN 60 mg/m2 (N=41) | IMGN 67.5 mg/m2 (N=4) | IMGN 75 mg/m2 (N=4)
Blood and Lymphatic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Endocrine (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (7) | 1 (1) | 0 (0)
Metabolism and Nutritional Disorders (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Surgical and Medical Procedures (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular Disorders (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General Disorders (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nervous System Disorders (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMGN 5 mg/m2 (N=4) | IMGN 10 mg/m2 (N=3) | IMGN 20 mg/m2 (N=4) | IMGN 40 mg/m2 (N=4) | IMGN 60 mg/m2 (N=41) | IMGN 67.5 mg/m2 (N=4) | IMGN 75 mg/m2 (N=4)
Blood and Lymphatic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (1)
cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (12) | 0 (0) | 1 (2)
Endocrine (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 4 (8) | 2 (4) | 1 (2) | 2 (6) | 32 (67) | 3 (5) | 4 (14)
General Disorders (General disorders) | 3 (4) | 1 (2) | 2 (2) | 2 (3) | 33 (61) | 3 (4) | 4 (4)
Hepatobiliary (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Immune System (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and Infestations (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 14 (17) | 1 (1) | 1 (2)
Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 0 (0)
Investigations (Investigations) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 18 (31) | 1 (1) | 1 (1)
Metabolism (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 1 (3) | 0 (0) | 17 (22) | 2 (2) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 21 (37) | 0 (0) | 1 (3)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 0 (0)
Nervous System (Nervous system disorders) | 1 (4) | 0 (0) | 0 (0) | 3 (4) | 31 (61) | 4 (7) | 3 (6)
Phychiatric (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 13 (18) | 0 (0) | 0 (0)
Renal and Urinary (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 9 (10) | 0 (0) | 0 (0)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 18 (26) | 1 (2) | 0 (0)
Skin and Subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 14 (20) | 1 (1) | 1 (1)
Vascular (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 8 (10) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No